CLINICAL TRIAL: NCT05247723
Title: Standard IV Cannula Aspiration (SIVCA): A Novel, Efficient and Minimally Invasive Testicular Sperm Aspiration Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Adham ZAAZAA, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIVCA
Record Dates: First submitted 2022-01-31; First posted 2022-02-21 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Non Obstructive Azoospermia
Keywords: Non Obstructive Azoospermia; Fine Needle Aspiration; Micro-TESE

STUDY DESIGN:
Intervention Model Description: On each patient, the testes were randomized to undergo testicular sperm aspiration using a standard IV cannula on one side, followed by surgical microscopic testicular sperm extraction on the contralateral testis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIVCA (Experimental): Aspirating testicular tissue using a standard IV cannula with applied negative pressure.
  Interventions: Procedure: Micro-TESE
- Micro-TESE (Active Comparator): Extracting testicular tissue surgically
  Interventions: Device: Standard IV Cannula for aspiration of testicular sperm

INTERVENTIONS:
Device: Standard IV Cannula for aspiration of testicular sperm — After local anesthesia, a wide bore 14-G standard IV cannula was introduced near the lower pole of the testis. The needle was withdrawn and the catheter introduced into the testicular tissue. A 20-ml syringe was secured to the catheter and constant negative pressure applied and secured with a clamp. Back and forth motions were performed covering as many areas of the testis as possible.
  Arms: Micro-TESE
Procedure: Micro-TESE — Conventional Microscopic Testicular Sperm Extraction (Micro-TESE), Open Testicular Biopsy using surgical Microscope
  Arms: SIVCA

SUMMARY:
Study question:

Can enough testicular tissue be aspirated for sperm retrieval in non-obstructive azoospermia (NOA), using a wide bore 14-G Standard IV cannula in comparison to micro-TESE?

Summary answer:

Standard IV cannula Aspiration (SIVCA) can yield an ample amount of testicular tissue sufficient for sperm retrieval through a single puncture site on the scrotum.

DETAILED DESCRIPTION:
What is known already:

The current conventional method of testicular sperm aspiration is fine needle aspiration (FNA). FNA has the advantage of being a cost-effective and minimally invasive procedure compared to open testicular sperm extraction (TESE). But FNA with its conventional 23-G needle may not always yield enough testicular tissue for sperm retrieval. Furthermore, FNA may require multiple punctures on the scrotum to retrieve enough tissues from different areas of the testis.

Study design, size, duration:

A 24 months prospective cohort study conducted at a specialized IVF center. A total of 130 men aged from 22 to 53 years old (35.03 +/- 9.04) with NOA and normal testicular volume (≥ 12ml) were enrolled in the study. The men had testicular biopsies taken at the day of their partners' ovum pick-up. On each patient, the testes were randomized to undergo SIVCA on one testis followed by micro-TESE on the contralateral testis.

Participants/materials, setting, methods:

After local anesthesia, a wide bore 14-G standard IV cannula was introduced near the lower pole of the testis. The needle was withdrawn and the catheter introduced into the testicular tissue. A 20-ml syringe was secured to the catheter and constant negative pressure applied and secured with a clamp. Back and forth motions were performed covering as many areas of the testis as possible. Micro-TESE was then performed on the contralateral testis.Sperm retrieval rates (SRR) will be compared between the two techniques using McNemar χ2 test. A P-value of less than 0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Non Obstructive Azoospermia
* Normal Sized testes (Above 12ml in volume)

Exclusion Criteria:

* Obstructive Azoospermia
* Small sized testes

Ages: 22 Years to 52 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 130 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Weight of Testicular Tissue Retrieval | Intraoperative
  If more than 0.3 grams of testicular tissue could be adequately collected from the procedure

SECONDARY OUTCOMES:
Sperm Retrieval Rate | Intraoperative
  If Sperm could be found in the collected testicular tissue sample, either aspirated or surgically extracted

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected during the trial after deidentification, beginning 9 months and ending 36 months after publication
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available upon reasonable request